CLINICAL TRIAL: NCT07338760
Title: Acute Effect of Core Stabilization Exercises Among Archers
Brief Title: The Acute Effects of Core Stabilization Exercises on Balance and Upper Extremity Functional Performance in Archers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AYŞE NUR ERTÜRK
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Archery; Core Stability; Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core training group (Experimental): The group that joins to core exercise training
  Interventions: Other: Core Training Exercise
- Control Group (No Intervention): The control group that performs any exercise

INTERVENTIONS:
Other: Core Training Exercise — Participants in the intervention group will perform a single session of core stabilization exercises targeting the deep and superficial trunk muscles. The exercise session will include static and dynamic stabilization exercises performed on stable and unstable surfaces, focusing on trunk control, postural alignment, and neuromuscular activation.
  Arms: Core training group

SUMMARY:
This randomized controlled study aims to investigate the acute effects of a single session of core stabilization exercises on balance and upper extremity functional performance in competitive archers. Core stability is essential for postural control, neuromuscular coordination, and efficient force transfer during archery shooting. Understanding the immediate effects of core stabilization exercises may support their use as an effective warm-up and performance-enhancing strategy in archery athletes.

DETAILED DESCRIPTION:
Archery is a precision sport requiring optimal postural stability, balance, and upper extremity control. Core muscles play a critical role in maintaining trunk stability and enabling effective force transmission along the kinetic chain. Insufficient core stability may negatively affect shooting accuracy, balance, reaction time, and upper extremity performance, while also increasing injury risk.

Although long-term effects of core stabilization exercises have been widely investigated, evidence regarding their acute effects on balance and upper extremity functional performance in archers is limited. This randomized controlled trial is designed to evaluate the immediate effects of a single session of core stabilization exercises added to routine warm-up on balance, upper extremity stability, reaction time, muscle strength, grip strength, and shooting performance.

Assessments will be conducted before and immediately after the intervention. The findings of this study may contribute to optimizing warm-up protocols and performance strategies in archery training and rehabilitation settings.

ELIGIBILITY:
Inclusion Criteria:

* Have been involved in licensed archery for at least 1 year

  * Be willing to participate in the program (both the athlete and their parent/guardian)
  * Be an athlete without any illness or disability that prevents participation in sports (as determined by a current medical report submitted to the club for licensing purposes)
  * Be able to read and write

Exclusion Criteria:

* ● Those with diagnosed mental or cognitive problems

  * Those who have undergone orthopedic surgery or received intra-articular steroid treatment within the last 6 months
  * Those with a diagnosed medical condition that could affect balance and shooting performance
  * Those with instability issues and associated joint movement restrictions
  * Those with acute muscle spasms and pain complaints
  * Those using painkillers, sedatives, alcohol, etc., or any other medication or substance that may affect shooting performance
  * Those with any diagnosis of injury related to the musculoskeletal system
  * Those actively involved in another sport besides archery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2025-08-09 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Lower extremity Balance Performance | Pre-intervention and immediately post-intervention
  Balance will be assessed using the Y Balance Test for lower extremities.

SECONDARY OUTCOMES:
Upper Extremity Functional Performance | Pre-intervention and immediately post-intervention
  Upper extremity functional performance will be evaluated using the Upper Quarter Y Balance Test.
Hand Reaction Time | Pre-intervention and immediately post-intervention
  Reaction time will be assessed using the BlazePod device.
Grip Strength | Pre-intervention and immediately post-intervention
  Grip strength will be measured using a digital hand dynamometer.
Shoulder Muscles Strengths | Pre-intervention and immediately post-intervention
  Shoulder muscles strengths will be measured using a hand-held dynamometer (MicroFET 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Hilal DENİZOĞLU KÜLLİ, Kağıthane, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No